CLINICAL TRIAL: NCT03462537
Title: Effect of Aerobic Exercise Associated With Abdominal Laser Therapy in Lipolytic Activity, Profile and Inflammatory Markers
Brief Title: Effect of Aerobic Exercise Associated With Abdominal Laser Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Andreia Noites, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AN-006
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Metabolic Disease
Keywords: Aerobic Exercise; Lipolytic Laser; Lipid Profile; C-reactive protein; Lipolysis
MeSH Terms: conditions — Metabolic Diseases | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group 1 (Experimental): This group performed aerobic exercise just after low level laser therapy in the abdominal region with eight electrodes distributed in line.
  Interventions: Device: Low level laser therapy; Device: Aerobic Exercise
- Experimental group 2 (Experimental): This group performed aerobic exercise just after low level laser therapy in the abdominal region with eight electrodes distributed in line, but low level laser therapy device was switched off.
  Interventions: Device: Aerobic Exercise; Device: Low level laser therapy without power
- Placebo group (Placebo Comparator): Low level laser therapy without power. This group performed the low level laser therapy protocol, but low level laser therapy device was switched off.
  Interventions: Device: Low level laser therapy without power

INTERVENTIONS:
Device: Low level laser therapy — Low level laser therapy protocol - The low level laser therapy protocol was performed in dorsal decubitus, with the head elevated at 45º. The electrodes were placed in line, in the abdominal region. The low level laser therapy device has a length of about 940nm, using 8 pads, which have 64 diodes, each one with 100mW. The duration of the application was established in 8 minutes.
  Arms: Experimental group 1
Device: Aerobic Exercise — Aerobic exercise protocol - 50 minutes of aerobic moderate-intensity exercise (45-55% of reserve heart rate) using Karvonen´s formula, performed on a cycloergometer. The duration of the exercise was divided into three parts: warm-up (from 0 to 5 minutes); body (from 5 to 45 minutes); and cooling (from 45 to 50 minutes). The entire protocol was monitored through the Polar® brand cardiofrequency and watch.
  Arms: Experimental group 1; Experimental group 2
Device: Low level laser therapy without power — Low level laser therapy protocol - The low level laser therapy protocol was performed in dorsal decubitus, with the head elevated at 45º. The electrodes were placed in line, in the abdominal region. The low level laser therapy device has a length of about 940nm, using 8 pads, which have 64 diodes, each one with 100mW. The duration of the application was established in 8 minutes. In this group low level laser therapy device was switched off.
  Arms: Experimental group 2; Placebo group

SUMMARY:
The purpose of the present study was to evaluate the effects of one session of aerobic exercise associated with low level laser therapy in lipolytic activity, lipid profile and inflammatory markers (C-reactive protein - CRP).

DETAILED DESCRIPTION:
The adipose tissue is the main energetic reserve, being constituted by adipocytes, cells that accumulate lipids inside its cytoplasm, in the form of triglycerides.

Fat deposition can occur both in the subcutaneous compartment and in the visceral compartment and is the result of a positive energy balance in which there is an imbalance between the amount of calories consumed and the amount of calories expended. Thus, an excess of energy storage occurs in the form of triglycerides in adipose tissue, which results from a sedentary lifestyle and a diet based on lipid rich nutrients. When fat deposition occurs in abdominal adipose tissue may favor the development of metabolic disorders.

Recently the effectiveness of an innovative physiotherapeutic intervention - low power laser therapy (LLLT) - on adipose tissue has been studied. This therapeutic modality stimulates cytochrome C oxidase, causing the release of nitric oxide, increased mitochondrial membrane potential and adenosine triphosphate (ATP) synthesis and the transient increase of reactive oxygen species (ROS). It is proposed that ROS creates temporary pores in the adipocyte membrane, allowing the release of its lipid content. It is also suggested that a regulation of cAMP occurs, which stimulates the lipolytic cascade, converting the triglycerides to fatty acids and glycerol. In this way, low level laser therapy seems to aid in the reduction of adiposity and in the decrease of cholesterol and triglycerides serum levels . In addition, it assists in the reduction of the inflammatory process related to obesity, by reducing the pro-inflammatory cytokines.

The aerobic exercise, due to its low-moderate intensity, enhances the stimulation of lipolysis, by decreasing plasma insulin concentration and elevating the level of catecholamines. In this way, it influences the lipid metabolism, seeming to improve the lipid profile, through the degradation of the triglycerides as energetic substrate. In addition, the regular practice of physical exercise seems to promote a decrease in the inflammation state due to metabolic changes, through the reduction of pro-inflammatory cytokines, namely interleukin-6 and, consequently, C-reactive protein.

The application of low level laser therapy in the abdominal region enhances the release of fat acids and glycerol into the bloodstream, increasing the availability of the substrate for muscle energy consumption. However, if they are not used as energy, free circulating fat acids may bind to glycerol and potentiate, again, the accumulation of triglycerides in abdominal adipocytes. Thus, aerobic exercise seems to be a good option in the fight against this re-esterification, since it is expected that the resulting fat acids will be converted to acetyl-CoA, entering the Krebs cycle, being used as energy source during aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 25 years.
* BMI between 18,5Kg/m2 and 29,9Kg/m2
* consider presenting abdominal fat

Exclusion Criteria:

* pregnant or intending to be in a period of 9 months
* participants with smoking habits
* participants with neoplasias, metabolic dysfunctions, renal pathologies, dermatological alterations
* participants with electronic devices
* participants with a condition that makes it impossible to practice physical exercise (disabling skeletal muscle pathologies and severe cardiorespiratory pathologies)
* participants under the effect of beta-blockers or other drugs which influence heart rate
* participants submitted to other fat reduce procedure

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-20 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Change in glycerol concentration | 10 minutes before the intervention and 5 minutes after the intervention
  Blood analysis collection was carried out with help from an clinical analysis technician.
Change in CRP concentration | 10 minutes before the intervention and 5 minutes after the intervention
  Blood analysis collection was carried out with help from an clinical analysis technician.
Change in lipid profile (LDL, HDL and triglyceride concentrations) | 10 minutes before the intervention and 5 minutes after the intervention
  Blood analysis collection was carried out with help from an clinical analysis technician.

REFERENCES:
- [Background] Afrooz PN, Pozner JN, DiBernardo BE. Noninvasive and minimally invasive techniques in body contouring. Clin Plast Surg. 2014 Oct;41(4):789-804. doi: 10.1016/j.cps.2014.07.006. PMID 25283463
- [Background] Ahmadian M, Wang Y, Sul HS. Lipolysis in adipocytes. Int J Biochem Cell Biol. 2010 May;42(5):555-9. doi: 10.1016/j.biocel.2009.12.009. Epub 2009 Dec 16. PMID 20025992
- [Background] Aquino Junior, A. E. (2012). Efeito do laser de baixa intensidade (830nm) associado ao exercício em ratos obesos exógenos. São Carlos: Universidade Federal de São Carlos
- [Background] Aquino AE Jr, Sene-Fiorese M, Castro CA, Duarte FO, Oishi JC, Santos GC, Silva KA, Fabrizzi F, Moraes G, Matheus SM, Duarte AC, Bagnato VS, Parizotto NA. Can low-level laser therapy when associated to exercise decrease adipocyte area? J Photochem Photobiol B. 2015 Aug;149:21-6. doi: 10.1016/j.jphotobiol.2015.04.033. Epub 2015 May 20. PMID 26026683
- [Background] Avci P, Gupta A, Sadasivam M, Vecchio D, Pam Z, Pam N, Hamblin MR. Low-level laser (light) therapy (LLLT) in skin: stimulating, healing, restoring. Semin Cutan Med Surg. 2013 Mar;32(1):41-52. PMID 24049929
- [Background] Avci P, Nyame TT, Gupta GK, Sadasivam M, Hamblin MR. Low-level laser therapy for fat layer reduction: a comprehensive review. Lasers Surg Med. 2013 Aug;45(6):349-57. doi: 10.1002/lsm.22153. Epub 2013 Jun 7. PMID 23749426
- [Background] Brown SA, Rohrich RJ, Kenkel J, Young VL, Hoopman J, Coimbra M. Effect of low-level laser therapy on abdominal adipocytes before lipoplasty procedures. Plast Reconstr Surg. 2004 May;113(6):1796-804; discussion 1805-6. doi: 10.1097/01.prs.0000117302.73214.1a. PMID 15114147
- [Background] da Silveira Campos RM, Damaso AR, Masquio DC, Aquino AE Jr, Sene-Fiorese M, Duarte FO, Tock L, Parizotto NA, Bagnato VS. Low-level laser therapy (LLLT) associated with aerobic plus resistance training to improve inflammatory biomarkers in obese adults. Lasers Med Sci. 2015 Jul;30(5):1553-63. doi: 10.1007/s10103-015-1759-9. Epub 2015 May 10. PMID 25958170
- [Background] Cavalheiro, C., Ferreira, A., & Assunção, F. (2012). O uso da eletrolipólise no tratamento da adiposidade localizada. Revisão integrativa. Ensaios e Ciência: Ciências Biológicas, Agrárias e da Saúde, 16(3), 157-165.
- [Background] Costa, A., Eberlin, S., Jorge, A., Mendonça, J., Kalies, A., & Pereira, C. (2014). Clinical study to assess abdominal circumferential reduction after treatment with lowfrequency. Surgical And Cosmetic Dermatology, 6(4), 320-324.
- [Background] Donges CE, Duffield R, Drinkwater EJ. Effects of resistance or aerobic exercise training on interleukin-6, C-reactive protein, and body composition. Med Sci Sports Exerc. 2010 Feb;42(2):304-13. doi: 10.1249/MSS.0b013e3181b117ca. PMID 20083961
- [Background] Elm CM, Wallander ID, Endrizzi B, Zelickson BD. Efficacy of a multiple diode laser system for body contouring. Lasers Surg Med. 2011 Feb;43(2):114-21. doi: 10.1002/lsm.21016. PMID 21384392
- [Background] de Ferranti S, Mozaffarian D. The perfect storm: obesity, adipocyte dysfunction, and metabolic consequences. Clin Chem. 2008 Jun;54(6):945-55. doi: 10.1373/clinchem.2007.100156. Epub 2008 Apr 24. PMID 18436717
- [Background] Glisezinski, & I. (2007). Mobilisation des lipides du tissu adipeux au cours de l'exercice physique. Science & Sports, 22(6), 280-285. doi:10.1016/j.scispo.2007.09.013
- [Background] Horowitz JF. Fatty acid mobilization from adipose tissue during exercise. Trends Endocrinol Metab. 2003 Oct;14(8):386-92. doi: 10.1016/s1043-2760(03)00143-7. PMID 14516937
- [Background] Jackson, R. F., Roche, G. C., & Wisler, K. (2010). Reduction in Cholesterol and Triglyceride Serum Levels Following Low-Level Laser Irradiation: A Noncontrolled, Nonrandomized Pilot Study. The American Journal of Cosmetic Surgery, 27, 177-184.
- [Background] Karu T. Photobiology of low-power laser effects. Health Phys. 1989 May;56(5):691-704. doi: 10.1097/00004032-198905000-00015. PMID 2651364
- [Background] Karu TI, Afanas'eva NI. [Cytochrome c oxidase as the primary photoacceptor upon laser exposure of cultured cells to visible and near IR-range light]. Dokl Akad Nauk. 1995 Jun;342(5):693-5. No abstract available. Russian. PMID 7670387
- [Background] Karu TI. Mitochondrial signaling in mammalian cells activated by red and near-IR radiation. Photochem Photobiol. 2008 Sep-Oct;84(5):1091-9. doi: 10.1111/j.1751-1097.2008.00394.x. Epub 2008 Jul 18. PMID 18651871
- [Background] Kennedy J, Verne S, Griffith R, Falto-Aizpurua L, Nouri K. Non-invasive subcutaneous fat reduction: a review. J Eur Acad Dermatol Venereol. 2015 Sep;29(9):1679-88. doi: 10.1111/jdv.12994. Epub 2015 Feb 9. PMID 25664493
- [Background] Lafontan M, Langin D. Lipolysis and lipid mobilization in human adipose tissue. Prog Lipid Res. 2009 Sep;48(5):275-97. doi: 10.1016/j.plipres.2009.05.001. Epub 2009 May 21. PMID 19464318
- [Background] Mulholland RS, Paul MD, Chalfoun C. Noninvasive body contouring with radiofrequency, ultrasound, cryolipolysis, and low-level laser therapy. Clin Plast Surg. 2011 Jul;38(3):503-20, vii-iii. doi: 10.1016/j.cps.2011.05.002. PMID 21824546
- [Background] Neira R, Arroyave J, Ramirez H, Ortiz CL, Solarte E, Sequeda F, Gutierrez MI. Fat liquefaction: effect of low-level laser energy on adipose tissue. Plast Reconstr Surg. 2002 Sep 1;110(3):912-22; discussion 923-5. doi: 10.1097/00006534-200209010-00030. PMID 12172159
- [Background] Nestor MS, Zarraga MB, Park H. Effect of 635nm Low-level Laser Therapy on Upper Arm Circumference Reduction: A Double-blind, Randomized, Sham-controlled Trial. J Clin Aesthet Dermatol. 2012 Feb;5(2):42-8. PMID 22468172
- [Background] Powers, S. K., & Howley, E. T. (2004). Fisiologia do Exercício - Teoria e Aplicação ao Condicionamento e ao Desempenho (5ª ed.). Brasil: Manole.
- [Background] Rosenbaum M, Prieto V, Hellmer J, Boschmann M, Krueger J, Leibel RL, Ship AG. An exploratory investigation of the morphology and biochemistry of cellulite. Plast Reconstr Surg. 1998 Jun;101(7):1934-9. doi: 10.1097/00006534-199806000-00025. PMID 9623840
- [Background] Stewart LK, Flynn MG, Campbell WW, Craig BA, Robinson JP, Timmerman KL, McFarlin BK, Coen PM, Talbert E. The influence of exercise training on inflammatory cytokines and C-reactive protein. Med Sci Sports Exerc. 2007 Oct;39(10):1714-9. doi: 10.1249/mss.0b013e31811ece1c. PMID 17909397
- [Background] Tafur J, Mills PJ. Low-intensity light therapy: exploring the role of redox mechanisms. Photomed Laser Surg. 2008 Aug;26(4):323-8. doi: 10.1089/pho.2007.2184. PMID 18665762